CLINICAL TRIAL: NCT00354731
Title: Clinical Efficacy of Pentoxifylline on Patients With Primary Nephrotic Syndrome
Brief Title: Efficacy of Pentoxifylline on Primary Nephrotic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 941103
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-10

CONDITIONS: Nephrotic Syndrome
Keywords: nephrotic syndrome, pentoxifylline, corticosteroid
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Pentoxifylline; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- corticosteroid (Active Comparator): Oral prednisolone (1 mg/kg/day) x 3 M, followed by gradual tapering (0.5 mg/kg/day at 6 M, 0.25 mg/day at 12 M, and discontinued at 18 M
  Interventions: Drug: Corticosteroid
- Pentoxifylline + corticosteroid (Experimental): Oral pentoxifylline 1,200 mg/day (for estimated GFR ≧60 ml/min) or 800 mg/day (estimated GFR 59-30 ml/min) x 6 months, followed by stepwise reduction (800 mg/day x 6 M, 400 mg/day x 6 M and discontinued at 18 M + oral prednisolone (1 mg/kg/day) x 3 M, followed by gradual tapering (0.5 mg/kg/day at 6 M, 0.25 mg/day at 12 M, and discontinued at 18 M
  Interventions: Drug: pentoxifylline; Drug: Corticosteroid

INTERVENTIONS:
Drug: pentoxifylline — Oral pentoxifylline 1,200 mg/day (for estimated GFR ≧60 ml/min) or 800 mg/day (estimated GFR 59-30 ml/min) x 6 months, followed by stepwise reduction (800 mg/day x 6 M, 400 mg/day x 6 M and discontinued at 18 M
  Other Names: Trental
  Arms: Pentoxifylline + corticosteroid
Drug: Corticosteroid — Oral prednisolone (1 mg/kg/day) x 3 M, followed by gradual tapering (0.5 mg/kg/day at 6 M, 0.25 mg/day at 12 M, and discontinued at 18 M
  Other Names: Predonin

SUMMARY:
We aim to investigate (1) the effects of combined pentoxifylline and corticosteroids, compared to that of corticosteroids, on patients with primary nephrotic syndrome; and if possible (2) the effects of pentoxifylline monotherapy on patients with primary nephrotic syndrome not suitable for or intolerant of standard corticosteroid therapy.

DETAILED DESCRIPTION:
Pentoxifylline (PTX) is a phosphodiesterase inhibitor that is used clinically to treat patients with peripheral vascular disorders. In addition to its hemorheologic activity, PTX possesses potent anti-inflammatory and immunomodulatory properties. In vivo, PTX has shown its ability to attenuate nephrotic syndrome secondary to membranous glomerulonephritis and lupus nephritis, and to reduce subnephrotic proteinuria of early and advanced diabetic nephropathy. However, the anti-proteinuric effect of PTX has been traditionally attributed to down-regulation of tumor necrosis factor (TNF)-alpha. Whether or not other inflammatory mediators are also affected by PTX has never been studied. Our previous works have shown that PTX can inhibit cytokine or albumin-induced monocyte chemoattractant protein (MCP)-1 production in vitro, and attenuate proteinuria in association with suppression of renal MCP-1 messenger ribonucleic acid expression in experimental glomerulonephritis. More recently, we have found that PTX lowers proteinuria by modulating renal MCP-1 production in a subgroup of human glomerular diseases. In this study, we aim to investigate whether combination of PTX and corticosteroids results in additive reduction in proteinuria, and higher remission rates in patients with primary nephrotic syndrome. The secondary objective is to study whether PTX monotherapy can be effective in patients with primary nephrotic syndrome not suitable for or intolerant of corticosteroid therapy.

This study is a prospective, open-labeled, comparative study including primary nephrotic patients randomized into 2 groups. Group A receives oral PTX plus oral prednisolone, whereas group B receives oral prednisolone alone. The active treatment duration is 1 year for both subgroups. The dose for PTX will be 1,200 mg/day (for estimated glomerular filtration rate (GFR) ≧60 ml/min) or 800 mg/day (estimated GFR 59-30 ml/min) x 6 months, followed by stepwise reduction (800 mg/day x 6 M, 400 mg/day x 6 M and discontinued at 18 M). The dose for prednisolone will be 1 mg/kg/day for the initial 3 months, then the dose will be gradually tapered, thus by 6 months the dose will be 0.5 mg/kg/day, and at 12 months the dose will be reduced to around 5-10 mg/day, and discontinued at 18 M. For patients not considered suitable for (eg., active chronic hepatitis B virus or hepatitis C virus infection), or intolerance of (eg., concomitant diabetes mellitus, active peptic ulcer disease) standard corticosteroid therapy, PTX 1,200 mg/day will be administered to them for a total of 1 year. Serum and urine specimens will be collected before initiation of therapy (day 0), and at month 1, 3, 6, and 12 after the commencement of therapy. GFR will be calculated by Cockcroft-Gault and simplified Modification of Diet in Renal Disease (MDRD) formula. Urinary protein excretion will be quantitated by spot urine protein/creatinine ratio. All biochemical and immunological analyses will be performed by the Department of Laboratory Medicine, National Taiwan University Hospital. Serum and urine samples will be measured for inflammatory mediators and podocyte markers by using commercial ELISA kits.

ELIGIBILITY:
Inclusion Criteria:

* biopsied-proved primary glomerular diseases, and nephrotic syndrome

Exclusion Criteria:

* History of allergy to pentoxifylline, Females are nursing or pregnant, Congestive heart failure (New York Heart Association functional class III or IV), Unstable angina, myocardial infarction, coronary artery bypass graft surgery, percutaneous coronary intervention, within the past 6 months prior to signing the informed consent form, Cerebral hemorrhage within the past 6 months prior to signing the informed consent form, Retinal hemorrhage within the past 6 months prior to signing the informed consent form, Known or suspected secondary hypertension, Uncontrolled hypertension with systolic blood pressure > 200 mmHg and/or diastolic blood pressure > 110 mmHg, Liver cirrhosis, Biliary obstructive disorders, Active malignancy or infection, Uncontrolled diabetes mellitus, GFR ≦ 30 ml/min/1.73 m2

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-08; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
changes from baseline in urinary protein excretion | 18 months

SECONDARY OUTCOMES:
change from baseline in creatinine and estimated GFR | 18 months

OTHER OUTCOMES:
Urinary nephrin, TNF-alpha and MCP-1 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Ming Chen, M.D., Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan